CLINICAL TRIAL: NCT01273090
Title: A Phase 1 Study of Imetelstat, a Telomerase Inhibitor, in Children With Refractory or Recurrent Solid Tumors and Lymphomas
Brief Title: Imetelstat Sodium in Treating Young Patients With Refractory or Recurrent Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL1112; COG-ADVL1112
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Brain and Central Nervous System Tumors; Lymphoma; Lymphoproliferative Disorder; Small Intestine Cancer; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific; recurrent childhood anaplastic large cell lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood brain stem glioma; recurrent childhood anaplastic astrocytoma; recurrent childhood anaplastic oligoastrocytoma; recurrent childhood anaplastic oligodendroglioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood diffuse astrocytoma; recurrent childhood fibrillary astrocytoma; recurrent childhood gemistocytic astrocytoma; recurrent childhood giant cell glioblastoma; recurrent childhood glioblastoma; recurrent childhood gliomatosis cerebri; recurrent childhood gliosarcoma; recurrent childhood oligoastrocytoma; recurrent childhood oligodendroglioma; recurrent childhood pilocytic astrocytoma; recurrent childhood pilomyxoid astrocytoma; recurrent childhood pleomorphic xanthoastrocytoma; recurrent childhood protoplasmic astrocytoma; recurrent childhood subependymal giant cell astrocytoma; recurrent childhood visual pathway and hypothalamic glioma; recurrent childhood visual pathway glioma; childhood pineal parenchymal tumor; recurrent childhood central nervous system embryonal tumor; childhood central nervous system choriocarcinoma; childhood central nervous system germ cell tumor; childhood central nervous system germinoma; childhood central nervous system mixed germ cell tumor; childhood central nervous system teratoma; childhood central nervous system yolk sac tumor; recurrent childhood pineoblastoma; childhood diffuse large cell lymphoma; childhood nasal type extranodal NK/T-cell lymphoma; childhood nodular lymphocyte predominant Hodgkin lymphoma; angioimmunoblastic T-cell lymphoma; childhood Burkitt lymphoma; childhood grade III lymphomatoid granulomatosis; childhood immunoblastic large cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; hepatosplenic T-cell lymphoma; intraocular lymphoma; noncutaneous extranodal lymphoma; peripheral T-cell lymphoma; post-transplant lymphoproliferative disorder; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; small intestine lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma; Lymphoproliferative Disorders; Lymphoma, Large-Cell, Anaplastic; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Recurrence; Astrocytoma; Oligodendroglioma; Glioblastoma; Neoplasms, Neuroepithelial; Optic Nerve Glioma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Extranodal NK-T-Cell; Hodgkin Disease; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — imetelstat

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: imetelstat sodium; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: imetelstat sodium
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Imetelstat sodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I clinical trial is studying the side effects and best dose of imetelstat sodium in treating young patients with refractory or recurrent solid tumors or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the maximum-tolerated dose (MTD) and/or recommended phase II dose of imetelstat sodium in children with refractory or recurrent solid tumors or lymphoma.
* To define and describe the toxicities of imetelstat sodium.
* To characterize the pharmacokinetics of imetelstat sodium in children with refractory or recurrent solid tumors or lymphoma.

Secondary

* To determine, in a preliminary manner, the antitumor effects of imetelstat sodium in children with refractory or recurrent solid tumors or lymphoma. (exploratory)
* To provide preliminary assessment of the biological activity of imetelstat sodium in children with recurrent or refractory malignancies by assessing telomerase activity, telomere length, hTERT protein, hTERT mRNA, and hTR levels in patient peripheral blood mononuclear cells (PBMNC) samples pretreatment and on treatment. (Exploratory)
* To assess telomerase activity, hTERT expression, telomere length, hTERT protein, hTERT mRNA, and hTR levels in patients' pretreatment tumor samples. (Exploratory)

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive imetelstat sodium IV over 2 hours on days 1 and 8. Treatment repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection at baseline and periodically during study for pharmacokinetic and correlative studies. Tumor tissue samples from diagnosis and/or subsequent tumor resections or biopsies may also be collected for correlative studies.

After completion of study therapy, patients are followed up for 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of refractory or recurrent solid tumors, including lymphoma

  * No CNS tumors or known CNS metastases (Part A, dose escalation)
  * CNS tumors or known CNS metastases allowed (Part B, maximum-tolerated dose or recommended phase II dose)

    * No prior or concurrent CNS hemorrhage on a baseline MRI within the past 14 days
  * All patients must have histologic verification of malignancy at original diagnosis or relapse except for:

    * Intrinsic brain stem tumors
    * Optic pathway gliomas
    * Pineal tumors and elevations of CSF or serum tumor markers including alpha-fetoprotein or beta-HCG
* Measurable or evaluable disease
* Disease for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood count criteria and they are not known to be refractory to red cell or platelet transfusions

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% (patients > 16 years of age) OR Lansky PS 50-100% (patients ≤ 16 years of age)
* ANC ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³ (transfusion-independent, defined as not receiving platelet transfusion within the past 7 days prior to enrollment)
* Creatinine clearance or radioisotope GFR ≥ 70 mL/min OR a serum creatinine based on age and/or gender as follows:

  * 0.6 mg/dL (1 to < 2 years of age)
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (≥ 16 years of age)
* Bilirubin (sum of conjugated and unconjugated) ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 110 U/L (ULN for ALT is 45 U/L)
* Serum albumin ≥ 2 g/dL
* aPTT < 1.2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use an effective contraception method
* No uncontrolled infection
* No patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

PRIOR CONCURRENT THERAPY:

* Recovered from acute toxic effects of all prior anti-cancer chemotherapy, immunotherapy, or radiotherapy
* At least 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosourea)
* At least 14 days since prior long-acting growth factor (e.g., Neulasta) or ≥ 7 days since prior short-acting growth factor
* At least 7 days since prior biologic or anti-neoplastic agent
* At least 6 weeks since any type of prior immunotherapy (e.g., tumor vaccines)
* At least 3 half-lives since last dose of a monoclonal antibody
* At least 2 weeks since prior local palliative radiotherapy (small port)

  * At least 24 weeks since prior total-body irradiation, craniospinal radiotherapy, or radiation to ≥ 50% of the pelvis
  * At least 6 weeks since prior substantial bone marrow radiation
* At least 12 weeks since prior transplantation or stem cell infusion with no evidence of active graft vs host disease
* Prior and concurrent stable or decreasing dose of corticosteroids within the past 7 days allowed
* No prior allogeneic transplant
* No other concurrent investigational drug
* No other concurrent anticancer agents including chemotherapy, radiotherapy, immunotherapy, or biologic therapy
* No concurrent cyclosporine, tacrolimus, or other agents to prevent either graft-versus-host disease post-bone marrow transplant or organ rejection post-transplant

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2011-05; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose and/or recommended phase II dose of imetelstat sodium in children with refractory or recurrent solid tumors or lymphoma | 21 Days
Toxicities of imetelstat sodium | Up to 30 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A. Thompson, MD, Principal Investigator — Baylor College of Medicine
Locations (23):
- United States (21):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Riley's Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec